CLINICAL TRIAL: NCT02133937
Title: A Single-center, Randomized Open-label, Single-dose, Parallel Group Study to Investigate the Relative Bioavailability of a High Concentration Liquid Formulation (Hclf) in Prefilled Syringes Versus the Reference Lyophilized Formulation (Lyof) of Gantenerumab Following Administration by Subcutaneous Injection in Healthy Volunteers
Brief Title: A Study Investigating the Bioavailability of a High Concentration Liquid Formulation Versus a Reference Lyophilized Formulation of Gantenerumab in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP29113
Record Dates: First submitted 2014-05-07; First posted 2014-05-08 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — gantenerumab

ARMS (2):
- High Concentration Liquid Formulation (HCLF) (Experimental)
  Interventions: Drug: gantenerumab
- Lyophilized formulation (Active Comparator)
  Interventions: Drug: gantenerumab

INTERVENTIONS:
Drug: gantenerumab — Single subcutaneous injection of a high concentration liquid formulation
  Arms: High Concentration Liquid Formulation (HCLF)
Drug: gantenerumab — Single subcutaneous injection of a lyophilized formulation
  Arms: Lyophilized formulation

SUMMARY:
This single-center, randomized open-label, single-dose, parallel group study will investigate the relative bioavailability of a high concentration liquid formulation (HCLF) versus the reference lyophilized formulation (LyoF) of gantenerumab. Healthy volunteers will be randomized 1:1 to receive single-dose gantenerumab by subcutaneous injection.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, 40 to 70 years of age inclusive. Healthy status is defined by absence of evidence any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, coagulation, serology and urinalysis. Some medical conditions are allowed that are well controlled by single stable medication
* A BMI between 18.0 to 30.0 kg/m2 inclusive
* Use of highly effective contraception until 6 months after study follow-up visit
* Agree not to donate blood or blood products for transfusion for the duration of the study and for one year after their dosing

Exclusion Criteria:

* Suspicion of alcohol or drugs abuse addiction using DSM IV criteria
* Regular smoker (> 5 cigarettes, > 1 pipeful or > 1 cigar per day), tobacco users and subjects on nicotine replacement therapy
* Prior administration of gantenerumab
* Participation in an investigational drug or device study within 60 days before dosing
* Donation of blood over 500 mL within three months before dosing
* Pregnancy or breast-feeding
* Any abnormal skin conditions or potentially obscuring tattoos, pigmentation or lesions in the area intended for subcutaneous injection
* Any familial history of early onset Alzheimer's disease
* Claustrophobia, presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, or foreign metal objects in the eyes, skin or body which would contraindicate an MRI scan

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of gantenerumab | Up to 13 weeks

SECONDARY OUTCOMES:
Incidence of adverse events | Approximately 21 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Lenexa, Kansas, United States